CLINICAL TRIAL: NCT02332434
Title: Effects of Various Bariatric Surgical Procedures on Intestinal Triglyceride-rich-lipoprotein (TRL) Metabolism in Obese Type 2 Diabetic Patients
Brief Title: Effects of Various Bariatric Surgical Procedures on Intestinal TRL Metabolism in Obese Type 2 Diabetic Patients
Acronym: MISTRAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-15; RCAPHM14_0179 (Registry Identifier: APHM)
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sleeve gastrectomy (Experimental): bariatric surgery procedure based exclusively on the gastric restriction (the sleeve gastrectomy).
  Interventions: Other: stable isotope enrichment methodology (5,5,5-D3-L-Leucine)
- gastric bypass (Experimental): bariatric surgery procedure associating a malabsorption (the gastric bypass).
  Interventions: Other: stable isotope enrichment methodology (5,5,5-D3-L-Leucine)

INTERVENTIONS:
Other: stable isotope enrichment methodology (5,5,5-D3-L-Leucine)

SUMMARY:
Rational: The world and french epidemic of obesity and diabetes represents a major problem of public health. The prevalence in France, in the adult population, is 15 % corresponding to 6.9 million people for obesity and 6 % corresponding to 3.9 million people for diabetes. Morbidly obesity (body mass index 40 kg/m²), the most serious, is more and more frequent. Cardiovascular diseases are the first cause of morbidity and mortality. The atherogenic dyslipidemia of these insulin-resistant obese type 2 diabetic patients characterized by the quartet: elevated plasma triglycerides, low high-density lipoprotein-cholesterol, increased proportion of small and dense low-density lipoproteins, is widely explained by the blood accumulation of TRL from the liver and the intestine, and represents a major cardiovascular risk factor. The overproduction of intestinal TRL (which apoprotein B48 is the specific tracer) is a constituent recently recognized of insulin-resistance and the atherogenous role of these intestinal TRL has been shown. In view of this important overmortality and the failures of the medical, nutritional, dietary and psychotherapeutic combined treatment, the bariatric surgery quickly developed. Two main procedures are performed: 1 based exclusively on the gastric restriction (the sleeve gastrectomy) and one associating a malabsorption (the gastric bypass).

Objectives: The main objective of this study is to compare the effect of each surgical procedure and the differential effect of the 2 bariatric surgery procedures on the production and clearance rates of the intestinal TRL. The secondary objectives are to compare the effect of each surgical procedure and the differential effect of the 2 bariatric surgery procedures on the production and clearance rates of the hepatic TRL and to document the potential links between the expected reduction of these productions after the surgery and the loss of weight, the improvement of the insulin-sensitivity, the changes in hormones, the decrease of the inflammatory state, the changes in energy expenditure, body composition and energy intake.

Methods: It is a multicentric, prospective, comparative study of cohorts. After identification of the eligible subjects, the kinetics (production and clearance rates) of intestinal and hepatic TRL will be performed in the hospital, using established stable isotope enrichment methodology (5,5,5-D3-L-Leucine), in 2 groups of obese patients (15 patients per surgery procedure), before and 6 months after the surgery.

Perspectives: A better understanding of the dyslipidemia of obese type 2 diabetic patients and the factors modulating this dyslipidemia may lead to develop new dietary and/or drugs and/or surgical treatments targeted at the enterocyte to improve the lipid profile of these patients and reduce the incidence of cardiovascular diseases. Moreover, a differential effect between the 2 surgical procedures could help to choose the best surgical procedure for obese type 2 diabetic patients depending on the lipid profile at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a body mass index between 35 and 60 kg / m²
* Subject with no contradiction to the 2 surgical techniques studied: Sleeve Gastrectomy and Gastric Bypass
* Subject with type 2 diabetes as defined
* Subject not having presented cardiovascular events (myocardial infarct, stroke, peripheral ischemia) in the previous 6 months

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
production and clearance rates of intestinal and hepatic TRL, in 2 groups of obese patients (15 patients per surgery procedure), before and 6 months after the surgery. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux Marseille
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, France

REFERENCES:
- [Derived] Frances L, Croyal M, Ruidavets JB, Maraninchi M, Combes G, Raffin J, de Souto Barreto P, Ferrieres J, Blaak EE, Perret B, Moro C, Valero R, Martinez LO, Viguerie N. Identification of circulating apolipoprotein M as a new determinant of insulin sensitivity and relationship with adiponectin. Int J Obes (Lond). 2024 Jul;48(7):973-980. doi: 10.1038/s41366-024-01510-w. Epub 2024 Mar 15. PMID 38491190